CLINICAL TRIAL: NCT07274540
Title: The Effects Of Front Arm Band Orthosis On Pain, Functionalite And Grip Force Evaluation To Person Of Play Instrument
Brief Title: Use Of Orthotics To Reduce Pain In Musicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Tuba YILDIZ, Lecturer, Medipol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.1378
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Musculoskeletal Pain; Overuse Syndrome; Tendinopathy, Elbow; Musculoskeletal Pain and Functional Impairment in Musicians
Keywords: Forearm Orthosis; Musician's Pain; Grip Strength; Evaluation; Instrument; Pain
MeSH Terms: conditions — Musculoskeletal Pain; Cumulative Trauma Disorders; Elbow Tendinopathy; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orthosis Group (Experimental): All participants received the Forearm Strap Orthosis intervention for a total period of 4 weeks. Measurements for primary and secondary outcomes were collected at baseline (pre-intervention) and immediately following the 4-week orthosis usage period (post-intervention). Data collection for this single-group intervention study was completed in 2020.
  Interventions: Device: Foream Band Orthosis

INTERVENTIONS:
Device: Foream Band Orthosis — The Forearm Band Orthosis was applied and used by participants for 4 weeks during instrumental music playing sessions and daily activities. The orthosis aimed to provide counterforce to the muscle tendon unit to reduce tension at the epicondyle and alleviate pain associated with repetitive strain.

SUMMARY:
This interventional clinical study investigates the effectiveness of applying a forearm strap orthosis in 30 individuals experiencing forearm pain due to playing a musical instrument. Participants used the orthosis for 4 weeks. The primary objective is to evaluate the changes in pain levels and grip strength following this period. The study also explores the potential of this intervention to improve functionality and quality of life.

DETAILED DESCRIPTION:
The therapeutic and biomechanical effects of orthoses are utilized in the management of musculoskeletal disorders frequently encountered in instrumental musicians; this interventional study aims to prospectively evaluate the effect of a standardized forearm strap orthosis intervention on pain intensity, grip strength, and upper extremity functionality after a 4-week usage period in instrumental musicians. The study employs an Interventional type, single-group assignment, non-randomized pre-post design, enrolling 30 individuals from the Sulukule Art Academy of Fatih Municipality who meet the inclusion criteria. The primary outcome measures are the McGill Melzack Pain Questionnaire and Visual Analogue Scale (VAS) scores, grip strength values measured with the Jamar dynamometer, and Disabilities of the Arm, Shoulder, and Hand (DASH-T) Questionnaire scores, all obtained pre- and post- orthosis use. The secondary outcome measure is the evaluation of quality of life using the Short Form 36 (SF-36) Quality of Life Survey.

ELIGIBILITY:
Inclusion Criteria:

* Participants were between 18 and 55 years old at the time of enrollment.
* Participants had been playing an instrument for more than six months.
* Participants had been playing an instrument for at least one hour a day.
* Participants were willing and able to adapt to orthotic treatment.

Exclusion Criteria:

* Participants had a history of surgery and/or trauma to the elbow where orthosis treatment was required.
* Participants were receiving physiotherapy treatment within the last 6 months.
* Participants had an acute injury that prevented performance.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain Intensity as Measured by the Visual Analog Scale (VAS) | Baseline and 4 weeks
  The VAS was a valid measure that recorded participants' perceived pain intensity. A decrease in the VAS score was evaluated. VAS ranges from a minimum of 0 (no pain) to a maximum of 10 (the most severe pain imaginable); higher scores indicate worse (more severe) pain.
Change from Baseline in Pain Experience Measured by the McGill Melzack Pain Questionnaire Score (MPQ-PRI) | Baseline and 4 weeks
  It was a questionnaire that measured the sensory, emotional, and evaluative aspects of pain. The decrease in the score was evaluated. The MPQ-PRI ranges from a minimum of 0 (no pain) to a maximum of 78 (the most severe and comprehensive pain); higher scores indicate a worse and more multidimensional pain experience.
Change from Baseline in Isometric Grip Strength using Jamar Dynamometer | Baseline and 4 weeks
  The maximum isometric grip strength of the affected hand was measured using the Jamar Dynamometer device.
Change from Baseline in Upper Extremity Functional Status using the Disabilities of the Arm, Shoulder, and Hand (DASH-T) Score | Baseline and 4 weeks
  It was a standardized questionnaire that measured upper extremity disability and its symptoms. A decrease in the DASH-T score (increased functionality) was evaluated.

SECONDARY OUTCOMES:
Change from Baseline in Quality of Life (SF-36) | Baseline and 4 weeks
  It was a survey that assessed the physical and mental components of quality of life. The increase in the SF-36 score was evaluated. The scores obtained from the form range from a minimum of 0 (poorest mental health and function) to a maximum of 100 (best function); higher scores indicate better physical and mental health and functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Yıldız, Lecturer, PhD student, Principal Investigator — Medipol University
Locations (1):
- Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. This decision is based on the informed consent provided by the participants, which did not grant permission for future data sharing beyond the scope of the original research project. Additionally, the study's sponsor does not possess the institutional infrastructure or dedicated resources required to de-identify, host, and manage a controlled data access platform for external investigators. The study results will be published in the scientific literature as aggregate data to ensure patient confidentiality and compliance with ethical approvals.